CLINICAL TRIAL: NCT05256524
Title: Is Anti-Factor Xa Associated With Mortality, Thromboembolism and Bleeding in Patients With Critical COVID-19 Patients on Low-Molecular-Weight Heparin?
Brief Title: Is Anti-Factor Xa Associated With Outcome in Patients With Critical COVID-19 on Low-Molecular-Weight Heparin?
Acronym: AntiXCOVID
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Lund University (Other)
Responsible Party: Principal Investigator, Sandra Jonmarker, Principal investigator, MD, PhD-student, Karolinska Institutet
Other Study IDs: AntiFactorXa in Covid-19
Record Dates: First submitted 2022-02-23; First posted 2022-02-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Covid19; Thromboembolism; Bleeding
Keywords: Low-molecular-weight Heparin; Anti-Factor Xa; Critical Care
MeSH Terms: conditions — COVID-19; Thromboembolism; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — anti-Factor Xa
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with critical COVID-19 responding to LMWH treatment: Responders are defined as patient who achieve aFXa-levels, peak or trough, within target-range as excepted from the given dose of LMWH.
  Interventions: Drug: The effect of LMWH; Diagnostic Test: Monitoring frequency of aFXa-levels
- Patients with critical COVID-19 not responding to LMWH treatment: Non-responders are defined as patients who do not achieve aFXa-levels, peak or trough, within target-range as excepted from the given dose of LMWH.
  Interventions: Drug: The effect of LMWH; Diagnostic Test: Monitoring frequency of aFXa-levels

INTERVENTIONS:
Drug: The effect of LMWH — Quantified by aFXa-levels
Diagnostic Test: Monitoring frequency of aFXa-levels — The frequency of aFXa-levels being sampled, analysed and integrated as a possible part of the basis for clinical decisionmaking

SUMMARY:
Patients with critical COVID-19 are hyper-coagulable and optimal thromboprophylaxis treatment differs with stage and severity. The most commonly used drug for thromboprophylaxis in the intensive care unit (ICU) is low-molecular-weight heparin (LMWH). In contrast to unfractionated heparins, the effects of LMWH usually do not require monitoring. Exceptions from this are when elimination of LMWH is impaired, extremes in age and weight, to identify deviations from predicted pharmacokinetics, and if there is an unexpected clinical response. The unexpected high incidence of thromboembolic complications among patients with critical COVID-19 compared to critically ill non-COVID-19 patients could motivate monitoring. The activity of LMWH is monitored by quantifying the presence of anti-Factor Xa (aFXa). The aim of this study is to investigate if the level and the monitoring frequency of aFXa is associated to mortality, thrombosis and bleeding in patients with critical COVID-19 treated with LMWH and therefore could be used as a potential tool to guide LMWH-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with critical COVID-19 and respiratory failure
* Positive SARS-CoV-2 test
* LMWH-effect monitored by aFXa, as a trough or peak value, after at least four doses at a twice daily regime

Exclusion Criteria:

* Diagnosed thromboembolism or major bleeding during their COVID-illness prior to ICU-admission or as a reason or contributing factor for the ICU-admission.
* Transferred to or from an ICU in other hospital/region making data collection regarding baseline data/outcomes not possible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with critical COVID-19 and respiratory failure admitted to ICU at Södersjukhuset, Karolinska Sjukhuset and Skånes Universitetssjukhus, in Sweden, between March 1 2020 and May 31 2021 are eligible.
  Patients will be included on their first admission to the ICU if admitted more than once. First admission can be replaced by the second one if the first one is considered very short/insignificant compared to the second one. If a patient is transferred from one ICU to another this will be considered the same admission but they will be grouped according to their initial ICU.
Sampling Method: Non-Probability Sample
Enrollment: 1520 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-08-29 (Actual)

PRIMARY OUTCOMES:
Mortality | 90 days from ICU admission
  90-day mortality

SECONDARY OUTCOMES:
Thromboembolic events | 28 days from ICU-admission
  Thromboembolic events are defined as the cumulative proportion of pulmonary embolism (PE), ischemic stroke and deep venous thrombosis (DVT).
  PE must be verified by computed tomography or by clinical suspicion as cause of deterioration combined with findings of acute strain of the right heart on echocardiography. Ischemic stroke must be verified by computed tomography. DVT must by verified by ultrasound or by computed tomography.
Bleeding events | 28 days from ICU-admission
  Bleeding events are categorized according to the World health organization (WHO) bleeding scale: 1) Petechiae, tissue hematoma, oropharyngeal bleeding, 2) Mild blood loss, hematemesis, macroscopic hematuria, hemoptysis, joint bleeding, 3) Gross blood loss requiring red blood cell transfusion and/or hemodynamic instability, 4) Debilitating blood loss, severe hemodynamic instability, fatal bleeding, or central nervous system bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Jonmarker, MD, Principal Investigator — Stockholm South General Hospital
Locations (1):
- Södersjukhuset, Stockholm, Sweden

REFERENCES:
- [Derived] Jonmarker S, Litorell J, Alarcon F, Al-Abani K, Bjorkman S, Farm M, Grip J, Soderberg M, Hollenberg J, Wahlin RR, Kander T, Rimling L, Martensson J, Joelsson-Alm E, Dahlberg M, Cronhjort M. A retrospective multicenter cohort study of the association between anti-Factor Xa values and death, thromboembolism, and bleeding in patients with critical COVID-19. Thromb J. 2023 Oct 2;21(1):101. doi: 10.1186/s12959-023-00541-z. PMID 37784131